CLINICAL TRIAL: NCT00418769
Title: A Randomized, Open Label, Two-arm, Three Period Crossover Bioavailability Study Comparing Two New Nilotinib Tablet Formulations to an Established Nilotinib Capsule Formulation in Healthy Volunteers
Brief Title: Bioavailability Study Comparing Two New Nilotinib Tablet Formulations to an Established Nilotinib Capsule Formulation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2117
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2012-04

CONDITIONS: Healthy
Keywords: nilotinib; bioavailability; tablet; capsule; PK; healthy, subject(s),
MeSH Terms: interventions — nilotinib

ARMS (2):
- Nilotinib Tablet Formulations (Experimental)
  Interventions: Drug: Nilotinib
- Established Nilotinib Capsule Formulation (Active Comparator)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib

SUMMARY:
Bioavailability study comparing two new nilotinib tablet formulations to an established nilotinib capsule formulation in healthy volunteers

ELIGIBILITY:
Inclusion

1. Healthy adult male (18 - 55 yrs) and sterile or post menopausal female subjects
2. Body weight must be ≥50 kg and <100 kg, with a body mass index (BMI) >18 but <33.
3. Laboratory parameter values must fall within the normal range

Exclusion

1. Female who is pregnant or breast feeding.
2. Contraindication to receiving nilotinib.
3. Smokers or user of tobacco products
4. A past medical history of clinically significant Electrocardiogram abnormalities, or a history/family history of long QT-interval syndrome.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-06; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
bioavailability of nilotinib

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

REFERENCES:
- See also: Results for CAMN107A2117 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2498